CLINICAL TRIAL: NCT00755196
Title: A Double-Blind, Randomized, 12 Week, Bilateral Study of the Safety and Efficacy of AN2728 Ointment, 5%, Versus Ointment Vehicle in the Treatment of Patients With Plaque Type Psoriasis
Brief Title: Safety and Efficacy Study of A Novel Ointment to Treat Plaque Type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AN2728-PSR-202; C3291015 (Other: Pfizer)
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Psoriasis
Keywords: Plaque Type Psoriasis; Topical
MeSH Terms: conditions — Psoriasis | interventions — crisaborole; Ointments

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): AN2728 Ointment, 5%
  Interventions: Drug: AN2728
- 2 (Placebo Comparator): AN2728 Ointment vehicle
  Interventions: Drug: Ointment vehicle

INTERVENTIONS:
Drug: AN2728 — AN2728 Ointment, 5%, twice daily for 12 weeks
  Other Names: AN2728 Ointment, 5%
  Arms: 1
Drug: Ointment vehicle — Ointment vehicle, twice daily for 12 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of AN2728 Ointment, 5%, compared to Ointment Vehicle, applied twice daily for 12 weeks, in the treatment of plaque type psoriasis

DETAILED DESCRIPTION:
This is a single center, randomized, double-blind, vehicle-controlled, bilateral design. Patients will apply both test articles, AN2728 Ointment, 5%, and Ointment Vehicle twice daily for 12 weeks. The assigned study medication will be applied to two comparable treatment targeted plaques identified at baseline. One test article will be applied to one plaque and the other test article to an anatomically distinct plaque. All efficacy evaluations will be measured from only the two plaques identified at the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >18 years of age at time of enrollment
2. The clinical diagnosis of stable plaque psoriasis
3. Two target plaques of similar severity

   * ≥ 5 cm2 but ≤ 100 cm2 computed by multiplying the greatest diameter of the plaque by the diameter of the plaque perpendicular to the greatest diameter
   * Bilaterally located (right/left) plaques on the arms or distinct plaques located on the trunk. Plaques located on the trunk must be separated by at least 10 cm and will be designated by the Investigator as either left/right or front/back or upper/lower
   * Overall target plaque severity score (OTPSS) of 2-4 (mild to moderate) with no more than a 1 point difference in the scores of the individual plaques
4. Normal or not clinically significant screening laboratory results
5. Willing and able to apply study drug as directed, comply with study instructions and commit to all follow-up visits
6. Ability to understand, agree to and sign the study Informed Consent Form (ICF) prior to initiation of any protocol related procedures

Exclusion Criteria:

1. Any dermatological conditions that could interfere with clinical evaluations or any disease state or physical condition which might expose the patient to an unacceptable risk by study participation
2. Any underlying disease(s) or other dermatological conditions that require the use of exclusionary topical or systemic therapy (see below).
3. Known sensitivity to any of the components of the study medication
4. Spontaneously improving or rapidly deteriorating psoriatic plaques or pustular/exfoliative, guttate, erythrodermic or other non-plaque form of psoriasis
5. Concomitant use of topical or systemic therapies that might alter the course of psoriasis
6. Females of child bearing potential. Females must be post-menopausal or surgically sterile (oophorectomy).
7. Washout periods of:

   * Topical drugs that might alter the course of psoriasis: 2 weeks
   * Oral retinoids: 8 weeks
   * Non-retinoid systemic drugs that might alter the course of psoriasis: 4 weeks
   * PUVA: 4 weeks
   * UVB therapy: 4 weeks
   * Use of emollients/moisturizers on area(s) to be treated: 2 days to baseline visit
8. AIDS or AIDS related illness
9. Concurrent participation in another drug research study or within 30 days of enrollment
10. Use of lithium or hydroxychloroquine containing products (i.e. Plaquenil)
11. Use of a beta-blocking medication (i.e. propranolol) if the dose has not been stabilized for at least 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- IMIC, Mexico City, Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Groups:
- AN2728 5 Percent (%) Ointment + Ointment Vehicle: AN2728 5 % ointment and ointment vehicle were applied to 2 comparable and anatomically distinct treatment-targeted plaques, respectively within each participant, twice daily for 12 weeks. Plaques were identified at Baseline (Day 1) by investigator.
Period: Overall Study
Arm/Group | AN2728 5 Percent (%) Ointment + Ointment Vehicle
Started | 30
Completed | 28
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficiency | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants who received the study medication.
Groups:
- AN2728 5% Ointment + Ointment Vehicle: AN2728 5 % ointment and ointment vehicle were applied to 2 comparable and anatomically distinct treatment-targeted plaques, respectively within each participant, twice daily for 12 weeks. Plaques were identified at Baseline (Day 1) by investigator.
Arm/Group | AN2728 5% Ointment + Ointment Vehicle
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (8.63)
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Lowering of Overall Target Plaque Severity Score (OTPSS) at Day 84
Description: OTPSS is a scale to assess plaque severity. Each target plaque was scored by the investigator on severity scale ranging from 0 (no plaque) to 8 (very severe plaque), where higher score indicated more severity of a plaque. In this outcome measure, percentage of participants with reduced OTPSS at Day 84 were reported and comparison of ointment and vehicle treated plaque was given as 'Ointment treated plaque versus (vs.) vehicle treated plaque' and 'Vehicle treated plaque vs. ointment treated plaque'.
Time Frame: Day 84
Population: ITT population included all randomized participants who received the study medication.
Measure: Number; unit: percentage of participants
Arm/Group | AN2728 5% Ointment + Ointment Vehicle
Number analyzed (Participants) | 30
percentage of participants
  Ointment treated plaque vs. vehicle treated plaque | 53.3
  Vehicle treated plaque vs. ointment treated plaque | 30.0
Statistical Analysis 1: Comparison: AN2728 5% Ointment + Ointment Vehicle; Test type: Superiority or Other; p = 0.23, 2-sided sign test

2. Secondary Outcome: Percentage of Participants With Lowering of Overall Target Plaque Severity Score (OTPSS) At Day 7, 14, 28, 42, 56, 70, 91
Description: OTPSS is a scale to assess plaque severity. Each target plaque was scored by the investigator on severity scale ranging from 0 (no plaque) to 8 (very severe plaque), where higher score indicated more severity of a plaque. In this outcome measure, percentage of participants with reduced OTPSS at Day 7, 14, 28, 42, 56, 70 and 91 were reported and comparison of ointment and vehicle treated plaque was given as 'Ointment treated plaque vs. vehicle treated plaque' and 'Vehicle treated plaque vs. ointment treated plaque'.
Time Frame: Day 7, 14, 28, 42, 56, 70, 91
Population: ITT population included all randomized participants who received the study medication.
Measure: Number; unit: percentage of participants
Groups:
- AN2728 5% Ointment + Ointment Vehicle: AN2728 5 % ointment and ointment vehicle were applied to 2 comparable and anatomically distinct treatment- targeted plaques, respectively within each participant, twice daily for 12 weeks. Plaques were identified at Baseline (Day 1) by investigator.
Arm/Group | AN2728 5% Ointment + Ointment Vehicle
Number analyzed (Participants) | 30
percentage of participants
  Day 7: Ointment treated vs.vehicle treated plaque | 10.0
  Day 7: Vehicle treated vs.ointment treated plaque | 10.0
  Day 14: Ointment treated vs.vehicle treated plaque | 43.3
  Day 14: Vehicle treated vs.ointment treated plaque | 10.0
  Day 28: Ointment treated vs.vehicle treated plaque | 60.0
  Day 28: Vehicle treated vs.ointment treated plaque | 3.3
  Day 42: Ointment treated vs.vehicle treated plaque | 60.0
  Day 42: Vehicle treated vs.ointment treated plaque | 6.7
  Day 56: Ointment treated vs.vehicle treated plaque | 60.0
  Day 56: Vehicle treated vs.ointment treated plaque | 16.7
  Day 70: Ointment treated vs.vehicle treated plaque | 56.7
  Day 70: Vehicle treated vs.ointment treated plaque | 23.3
  Day 91: Ointment treated vs.vehicle treated plaque | 40.0
  Day 91: Vehicle treated vs.ointment treated plaque | 30.0

ADVERSE EVENTS:
Description: Same event may appear as both an Adverse Event (AE) and Serious Adverse Event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non serious in another participant, or 1 participant may have experienced both a serious and non serious event during the study. Safety population included all participants who used the study medication and provided a safety evaluation.
Arm/Group | AN2728 5% Ointment + Ointment Vehicle
Serious Adverse Events (participants affected / at risk) | 1/29
Other Adverse Events (participants affected / at risk) | 8/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AN2728 5% Ointment + Ointment Vehicle (N=29)
Drug eruption (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AN2728 5% Ointment + Ointment Vehicle (N=29)
Pharyngitis (Infections and infestations) | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 7
Scab (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.